CLINICAL TRIAL: NCT06073678
Title: Photobiomodulation in Gingival Graft Donor Areas: Clinical, Somatosensory, and Quality of Life Evaluations
Brief Title: Photobiomodulation in Palate Wounds: Somatosensorial Evaluation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Carla Andreotti Damante, Associate professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Photobiomodulation in palate
Record Dates: First submitted 2023-09-25; First posted 2023-10-10 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Surgical Wound
MeSH Terms: conditions — Surgical Wound | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will be masked by using a sham laser. Outcomes assessor will not be able to identify the experimental groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Photobiomodulation (Experimental): Red laser irradiation on palate wound at the day of the surgery and after 2, 4 and 6 days postoperatively. Protection of wound with surgical dressing during 7 days.
  Interventions: Other: Photobiomodulation
- Control (Active Comparator): Protection of wound with surgical dressing during 7 days.
  Interventions: Other: Protection with surgical dressing

INTERVENTIONS:
Other: Photobiomodulation — Irradiation with red laser on palate wound each 48h for 4 sessions.
  Other Names: Low level laser treatment; Low intensity laser treatment
  Arms: Photobiomodulation
Other: Protection with surgical dressing — Protection of the palatal wound with surgical dressing for 7 days
  Other Names: Protection of wound
  Arms: Control

SUMMARY:
The goal of this clinical trial is to compare the effects of photobiomodulation with red laser on gingival graft donor areas of the palate in comparison to only protection with wound dressing. The main questions it aims to answer are: Does photobiomodulation on the palate promote faster somatosensory recovery? Does photobiomodulation reduce pain in palate donor sites, improving the quality of life? Participants who need gingival graft surgeries will receive laser irradiation on the palate donor area or just protection with wound dressing. Data will be collected up to 60 days. Researchers will compare protection on the palate and protection plus laser irradiation to see if laser therapy may reduce pain and accelerate somatosensory normalization. Moreover, they will measure changes in the quality of life after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Palate with normal and healthy mucosa
* Patient with indication of gingival graft surgery

Exclusion Criteria:

* Patients using prosthesis with palate coverage
* Former removal of gingival graft in the palate
* Smokers
* Pregnancy and breastfeeding mothers
* Use of anticonvulsants and immunosuppressors

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Somatosensory recovery | 30 and 60 days postoperatively
  Mechanical and pain detection threshold measured with Von Frey filaments

SECONDARY OUTCOMES:
Assessment of Pain | 24 hours, 3 days, 7 days and 14 days
  Numeric analogue scale from zero to ten. Patients marks zero for no pain and ten for the worse pain.
Measurement of Quality of life | Baseline, 7 days and 14 days postoperatively
  Patients fill the Oral Health Impact Profile (OHIP-14) questionnaire. It comprises 14 questions about oral health problems. In each question the patient may answer if they he have those problems very often (coded 4), fairly often (coded 3), occasionally (coded 2), hardly ever (coded 1) or never (coded 0). Questionnaire scale ranges from 0 to 56 with higher scores indicating poorer quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Bauru School of Dentistry, Bauru, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhao H, Hu J, Zhao L. The effect of low-level laser therapy as an adjunct to periodontal surgery in the management of postoperative pain and wound healing: a systematic review and meta-analysis. Lasers Med Sci. 2021 Feb;36(1):175-187. doi: 10.1007/s10103-020-03072-5. Epub 2020 Jul 1. PMID 32613416
- [Background] Dias SB, Fonseca MV, Dos Santos NC, Mathias IF, Martinho FC, Junior MS, Jardini MA, Santamaria MP. Effect of GaAIAs low-level laser therapy on the healing of human palate mucosa after connective tissue graft harvesting: randomized clinical trial. Lasers Med Sci. 2015 Aug;30(6):1695-702. doi: 10.1007/s10103-014-1685-2. Epub 2014 Nov 6. PMID 25373688